CLINICAL TRIAL: NCT03271554
Title: Treatment Registry of Alecensa in Korean Patients With Anaplastic Lymphoma Kinase (ALK)-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Treatment Registry of Alectinib in Anaplastic Lymphoma Kinase (ALK)-Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer in Korea
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30132
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alectinib: Participants with ALK-positive, locally advanced or metastatic non-small cell lung cancer, who are treated with alectinib in accordance with local clinical practice and local labeling, are observed in this study.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — According to local labeling the recommended dose of alectinib is 600 mg given orally, twice daily with food (total daily dose of 1200 mg).
  Other Names: Alecensa

SUMMARY:
Alectinib was approved by the Ministry of Food and Drug Safety (MFDS) in Korea in Oct 2016. The purpose of this registry is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and effectiveness of the new drug so that the regulatory authority can manage the marketing approval properly.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who are administered alectinib at physician's discretion and fall into the approved indication in Korea.

Exclusion Criteria:

* Hypersensitivity to alectinib or any ingredient of alectinib;
* Pregnant or lactating women;
* Pediatric subjects (age </=18 years);
* Due to the presence of lactose, subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take alectinib.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ALK-positive, locally advance or metastatic non-small cell lung cancer, who are administered alectinib at physician's discretion in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 3 years
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. All AE events will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 3 years
  ORR will be determined according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 as assessed by physicians under routine clinical practice. Overall response rate was defined as the percentage of participants who had any evidence of Complete Response (CR) or Partial Response (PR): CR is defined as the disappearance of all target lesions and all nodes with short axis <10 millimeter (mm); PR is defined as >/=30% decrease in the sum of the longest diameter of target lesions. Target lesions are those lesions with longest diameter >/=10 mm and limits that are sufficiently well defined for their measurement to be considered reliable. Lymph nodes are target lesions if short-axis measures >/=15 mm. Maximum number of selected target lesions is 5 per participant and 2 per organ. Overall Response (OR) = CR + PR.
Complete Response (CR) | Up to approximately 3 years
  CR will be determined according to RECIST v1,1 as assessed by physicians under routine clinical practice and is defined as disappearance of all target lesions and all nodes with short axis <10 mm. Target lesions are those lesions with longest diameter >/=10 mm and limits that are sufficiently well defined for their measurement to be considered reliable. Lymph nodes are target lesions if short-axis measures >/=15 mm. Maximum number of selected target lesions is 5 per participant and 2 per organ.
Percentage of Participants with Partial Response (PR) | Up to approximately 3 years
  PR will be determined according to RECIST v1.1 as assessed by physicians under routine clinical practice and is defined as >/=30% decrease in the sum of the longest diameter of target lesions. Target lesions are those lesions with longest diameter >/=10 mm and limits that are sufficiently well defined for their measurement to be considered reliable. Lymph nodes are target lesions if short-axis measures >/=15 mm. Maximum number of selected target lesions is 5 per participant and 2 per organ.
Percentage of Participants with Stable Disease (SD) | Up to approximately 3 years
  SD will be determined according to RECIST v1.1 as assessed by physicians under routine clinical practice and is defined as neither response nor progression. Response is defined as at least >/=30% decrease in the sum of the longest diameter of target lesions. Progression is defined as >/= 20% increase in the sum of target lesions taking as reference the smallest sum measured during follow-up and >/= 5 mm in absolute value. Target lesions are those lesions with longest diameter >/=10 mm and limits that are sufficiently well defined for their measurement to be considered reliable. Lymph nodes are target lesions if short-axis measures >/=15 mm. Maximum number of selected target lesions is 5 per participant and 2 per organ.
Percentage of Participants with Progressive Disease (PD) | Up to approximately 3 years
  PD will be determined according to RECIST v1.1 as assessed by physicians under routine clinical practice and is defined as >/=20% increase in the sum of target lesions taking as reference the smallest sum measured during follow-up and >/= 5 mm in absolute value. Target lesions are those lesions with longest diameter >/=10 mm and limits that are sufficiently well defined for their measurement to be considered reliable. Lymph nodes are target lesions if short-axis measures >/=15 mm. Maximum number of selected target lesions is 5 per participant and 2 per organ.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- South Korea (37):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Dongnam Institute of Radiological & Medical Sciences, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Bucheon St Mary's hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Catholic Univ. of Incheon St.Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Inje University, Sanggye-Paik Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Severance Hospital, Seoul
  - Gangdong Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Soon Chun Hyang University Hospital; Department of Pulmonology and Allergy, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju